CLINICAL TRIAL: NCT03630094
Title: A Phase 1, Multiple-Dose, Open-Label Study to Determine and Compare Plasma and Intrapulmonary Concentrations of WCK 5222 (Cefepime and Zidebactam) in Healthy Adult Human Subjects
Brief Title: Plasma and Intrapulmonary Concentrations Study of WCK 5222
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Wockhardt (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: W-5222-104
Record Dates: First submitted 2017-03-17; First posted 2018-08-14 (Actual); Last update posted 2018-08-14 (Actual); Status verified 2018-08

CONDITIONS: PHA1A

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- FEP-ZID via intravenous (Experimental): total of 7 doses of FEP-ZID via intravenous infusion over 60 min at q8hr dosing regimen
  Interventions: Drug: FEP-ZID

INTERVENTIONS:
Drug: FEP-ZID — A total of 7 doses of FEP-ZID via intravenous infusion over 60 min at q8hr dosing regimen

SUMMARY:
This is a Phase 1, multiple dose, open-label pharmacokinetic study in healthy adult male and female subjects.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) greater than or equal to18.5 and less than or equal to 30 (kg per m2) and weight between 55.0 and 100.0 kg (both inclusive).
* Medical history without any major pathology as judged by the Investigator.
* Forced expiratory volume in 1 second (FEV1) of at least 70% of predicted value at screening.

Exclusion Criteria:

* History or presence of significant oncologic, cardiovascular, pulmonary, hepatic, renal, hematological, gastrointestinal,endocrine, immunologic, dermatologic, neurological, or psychiatric disease.
* Positive alcohol breath test or urine drug screen test at screening or confinement.
* Current use or has used tobacco or nicotine containing products 6 month prior to screening.
* Positive testing for HIV, Hepatitis B or Hepatitis C.
* History or presence of alcohol or drug abuse within the 2 years prior to screening.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2017-03-31 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2017-07-30 (Actual)

PRIMARY OUTCOMES:
concentrations of cefepime (FEP) and zidebactam in epithelial lining fluid (ELF) | Day 3
concentrations of cefepime (FEP) and zidebactam in alveolar macrophage (AM) | Day 3

SECONDARY OUTCOMES:
Number of adverse event reported | Day 3
number variation noted in 12-lead electrocardiogram | Day 3

CONTACTS AND LOCATIONS:
Locations (1):
- Pulmonary Associates, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: No